CLINICAL TRIAL: NCT05244356
Title: Effective Public Health Communication to Influence COVID-19 Vaccination Intent and Message Propagation: A Randomized Controlled Experiment
Brief Title: Health Communication to Influence COVID-19 Vaccination Intent and Message Propagation
Acronym: CONVINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: Institute for Health Behavioral Research, Malaysia (Unknown); University of Malaya (Other); UNICEF Malaysia (Unknown); Ministry of Health, Malaysia (Other Government); London School of Economics and Political Science (Other)
Responsible Party: Principal Investigator, Nicholas Hing Yee Liang, Researcher, Principle Investigator, Pharmacist, Clinical Research Centre, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NMRR-21-26-58107
Record Dates: First submitted 2022-02-10; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Respiratory Disease; Vaccine Refusal; Infectious Disease; Coronavirus Infections; Behavior, Health; Pneumonia; Respiratory Tract Infections; Lung Diseases; Pneumonia, Viral
Keywords: message; messaging; propagation; intent; vaccine; recommend
MeSH Terms: conditions — COVID-19; Respiration Disorders; Vaccination Refusal; Communicable Diseases; Coronavirus Infections; Health Behavior; Pneumonia; Respiratory Tract Infections; Lung Diseases; Pneumonia, Viral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Descriptive Norm (70%) (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing that about 70% of Malaysians have expressed acceptance for the COVID-19 vaccine.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Descriptive Norm (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing that the COVID-19 vaccine has been widely tested including with the elderly and people with existing health conditions, while subsequently highlighting that the vaccine was already received by millions worldwide.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Healthcare worker (HCW) recommendation (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content highlights recommendation from Malaysian healthcare workers to get the vaccine, since majority of them has already received it, including the Malaysian Health Director General
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Negative attribute framing (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing the rate of side effects occurring with COVID-19 vaccination in a negative frame.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Positive attribute framing (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing the rate of side effects occurring with COVID-19 vaccination in a positive frame.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Risky choice framing (Safety) (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing a risky choice frame which compares the death rates occurring with COVID-19 vaccination versus contracting the virus itself.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Risky choice framing (Side effects) (Experimental): Intervention in the form of a message likened to a social media post. Composed of 3 parts:
  1. Opening tag line highlighting the main concern that Malaysians have about the COVID-19 vaccine (safety and side effects)
  2. Message content describing a risky choice frame that compares the incidence rates of blood clots occurring with COVID-19 vaccination versus contracting COVID-19.
  3. Rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Control message (Experimental): Control message containing only rally slogan: "It's safe and effective!"
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + Descriptive Norm (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + HCW recommendation (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + Negative attribute framing (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + Positive attribute framing (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + Risky choice framing (Safety) (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure
- Combination message: Descriptive Norm (70%) + Risky choice framing (Side effects) (Experimental): Participants received 2 messages which were exposed one at a time. Sequence of message appearing randomly rotated.
  Interventions: Behavioral: Health message exposure

INTERVENTIONS:
Behavioral: Health message exposure — Participants exposed to a health message and requested to read it completely. Subsequently requested to answer post intervention questions that form basis for outcome measures.

SUMMARY:
This is a randomised controlled experiment in the form of a web based survey study which randomly exposes participants to different forms of public health messages, after which participants will be assessed on their intent to take up the COVID-19 vaccine, recommend the vaccine, and also willingness to propagate the exposed message.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the trial
* Malaysian nationality.
* Can understand either the English or Malay language.
* Aged 18 years or above

Exclusion Criteria:

* Received at least one COVID-19 vaccination dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5784 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Change in intent to accept the COVID-19 vaccine amongst the Malaysian adult population. | Immediately before and after message exposure during questionnaire administration.
  Outcome measure was assessed using a questionnaire answered through a 4 point ordinal scale. Scale ranges from '"Definitely no", "Not sure, but probably no", "Not sure, but probably yes"to Definitely yes".
Change in intent to recommend the COVID-19 vaccine to healthy adults. | Immediately before and after message exposure during questionnaire administration.
  Outcome measure was assessed using a questionnaire answered through a 5 point ordinal scale. Scale ranges from "Strongly disagree", "Disagree", "Not sure", "Agree", and "Strongly agree".
Change in intent to recommend the COVID-19 vaccine to elderly. | Immediately before and after message exposure during questionnaire administration.
  Outcome measure was assessed using a questionnaire answered through a 5 point ordinal scale. Scale ranges from "Strongly disagree", "Disagree", "Not sure", "Agree", and "Strongly agree".
Change in intent to recommend the COVID-19 vaccine to people with existing health conditions. | Immediately before and after message exposure during questionnaire administration.
  Outcome measure was assessed using a questionnaire answered through a 5 point ordinal scale. Scale ranges from "Strongly disagree", "Disagree", "Not sure", "Agree", and "Strongly agree".
Intent to share message on social media platform. | Immediately after message exposure during questionnaire administration.
  Outcome measure was assessed using a questionnaire answered through a 5 point ordinal scale.Scale ranges from "Strongly disagree", "Disagree", "Not sure", "Agree", and "Strongly agree".

SECONDARY OUTCOMES:
Moderators of vaccination intent. | Immediately after message exposure during questionnaire administration.
  Outcome measure assessed using a series of questions answered through a 5 point ordinal scale. Scale ranges from "Strongly disagree", "Disagree", "Not sure", "Agree", and "Strongly agree".
Reliability of various information sources about COVID-19. | Immediately after message exposure during questionnaire administration.
  Outcome measure assessed using a questionnaire that list out various types of information sources and having participants to rate the reliability for each source using a 5 point ordinal scale. Scale ranges from "Strongly not reliable", "Not reliable, "Not sure", "Reliable", and "Strongly reliable".

CONTACTS AND LOCATIONS:
Overall Officials: Yee Liang Hing, MSc., Principal Investigator — Clinical Research Centre, Malaysia
Locations (1):
- Institute for Clinical Research, National Institutes of Health, Malaysia, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hing NYL, Woon YL, Lee YK, Kim HJ, Lothfi NM, Wong E, Perialathan K, Ahmad Sanusi NH, Isa A, Leong CT, Costa-Font J. When do persuasive messages on vaccine safety steer COVID-19 vaccine acceptance and recommendations? Behavioural insights from a randomised controlled experiment in Malaysia. BMJ Glob Health. 2022 Jul;7(7):e009250. doi: 10.1136/bmjgh-2022-009250. PMID 35906015